CLINICAL TRIAL: NCT05613634
Title: Effect of Repetitive Transcranial Magnetic Stimulation on Vestibular Function and Self-rated Functional Recovery in Patients With Peripheral Vestibular Dysfunction
Brief Title: Effect of Repetitive Transcranial Magnetic Stimulation in Patients With Peripheral Vestibular Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Hosam Magdy Metwally, Hosam.Magdy.PT@o6u.edu.eg, October 6 University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 152947
Record Dates: First submitted 2022-11-06; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Peripheral Vestibular Dysfunction
Keywords: Vestibular dysfunction, repetitive transcranial magnetic stimulation, vestibular physical therapy exercises, vertigo, Activities of daily living.
MeSH Terms: conditions — Vertigo | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The study group received rTMS in addition to the vestibular physical therapy exercises
  Interventions: Device: Repetitive transcranial magnetic stimulation; Other: Cawthorne Cooksey exercises
- Control group (Experimental): Patients in control group received the vestibular physical therapy exercises, three sessions a week for four weeks
  Interventions: Other: Cawthorne Cooksey exercises

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — A high frequency (10 Hz) rTMs on the dominant dorsolateral prefrontal cortex (DLPFC) was applied with the Magstim Rapid Magnetic Stimulator, Magstim Company. Patients were seated in a chair, arms and legs relaxed, head stable, and no movement was allowed during the procedure. Motor threshold (MT) was determined before each session and was defined as the percent intensity output of the stimulator that generated a 50µV motor evoked response in the abductor pollicis brevis (APB) muscle in five out of 10 trials. The DLPFC of dominant hemisphere was localized on the scalp 5.5 cm anterior to the hot spot for the contralateral APB muscle along the parasagittal plane. The average MT was 50 % (range, 45-55%) of the maximal output of the stimulator. The initial mapping procedure was completed with the coil oriented at 45° lateral diagonal orientation roughly perpendicular to the central sulcus and the center of the coil applied tangentially to the scalp.
  Arms: Study group
Other: Cawthorne Cooksey exercises — Cawthorne Cooksey exercises were carried in the following sequence: First, bed exercises; eye movements (up and down, side to side, focusing on a finger that is one feet distance); head movements (bending up and down, side to side first with eye opened then closed). Second, sitting exercises involved same eye and head movements, shoulder shrugging, turning head and trunk alternately to the right and left, bending head and trunk forward, and pick an object from the ground. Third, standing exercises involved same eye, head, and shoulder movements, changing position from sitting to standing with eye open then closed, throw a ball from hand to hand above eye level, throw a ball from hand to hand beneath knee, changing position from sitting to standing and turn around in between. Fourth, moving around exercises where the patient revolved around a person sitting in the center who throw him a ball and to whom it was returned.

SUMMARY:
Background: Vestibular dysfunctions are common disorders in the adult population that can develop at any life decade. Most of the patients with vestibular dysfunction suffer from balance disorders and vertigo that may have a negative impact on daily living activities and social participation.

Objectives: To investigate the effect of repetitive transcranial magnetic stimulation added to vestibular physical therapy exercises on functional recovery in patients with vestibular dysfunction.

Hypothesis: There is no effect of repetitive transcranial magnetic stimulation added to vestibular physical therapy exercises on functional recovery in patients with vestibular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed by an audiologist with a chronic uncompensated unilateral peripheral vestibular weakness
* age ranged from 30 to 60 years, and duration of illness ranged from 4 to 32 months

Exclusion Criteria:

* benign paroxysmal positional vertigo
* bilateral peripheral vestibular weakness
* central vestibular disorders
* acute vestibular weakness
* vertigo of vascular origin (Vertebrobasilar insufficiency) or cervical origin

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Video-nystagmography (VNG) | 35 minutes
  The VNG was used to assess unilateral vestibular canal weakness. It was used with caloric testing to analyze eye movements using video imaging technology, in which hi-tech video goggles with infrared cameras were used

SECONDARY OUTCOMES:
Dizziness handicap inventory (DHI) | 20 minutes
  is used in clinical work and in research to assess the impact of dizziness on QoL. The self-report questionnaire was designed to quantify the handicapping effect of dizziness imposed by vestibular system disease. The Arabic version of the DHI has good validity and reliability for assessing patients' self-perception of the handicap and its impact on their QoL

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided